CLINICAL TRIAL: NCT06816992
Title: Phase 1b Study of ORIC-114 in Combination with Amivantamab in Patients with EGFR Exon20 Insertion Mutant NSCLC
Brief Title: ORIC-114 in Combination with Subcutaneous Amivantamab in Patients with EGFR Exon20 Insertion Mutant NSCLC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ORIC Pharmaceuticals (Industry)
Collaborators: Janssen Research and Development LLC (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ORIC-114-05
Record Dates: First submitted 2025-02-03; First posted 2025-02-10 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-02

CONDITIONS: Solid Tumors; EGFR Exon 20 Insertion Mutations; NSCLC; EGFR-mutated NSCLC
Keywords: NSCLC; EGFR mutations; EGFR exon20; EGFR exon 20 insertion mutations; ORIC-114; Amivantamab
MeSH Terms: interventions — amivantamab

STUDY DESIGN:
Intervention Model Description: Interval 3+3 dose escalation design followed by dose expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part 1 Dose Escalation level 1 (Experimental): ORIC-114 + amivantamab
  Interventions: Drug: ORIC-114 Dose 1 + amivantamab
- Part 1 Dose Escalation level 2 (Experimental): ORIC-114 + amivantamab
  Interventions: Drug: ORIC-114 Dose 2 + amivantamab
- Part 1 Dose Escalation level 3 (Experimental): ORIC-114 + amivantamab
  Interventions: Drug: ORIC-114 Dose 3 + amivantamab
- Part 2 Dose Expansion (Experimental): Two potential ORIC-114 dose levels + amivantamab
  Interventions: Drug: ORIC-114 Dose 2 + amivantamab; Drug: ORIC-114 Dose 3 + amivantamab

INTERVENTIONS:
Drug: ORIC-114 Dose 1 + amivantamab — ORIC-114 oral daily, amivantamab subcutaneous weekly for 4 weeks followed by every 4 week injection
  Arms: Part 1 Dose Escalation level 1
Drug: ORIC-114 Dose 2 + amivantamab — ORIC-114 oral daily, amivantamab subcutaneous weekly for 4 weeks followed by every 4 week injection
  Arms: Part 1 Dose Escalation level 2; Part 2 Dose Expansion
Drug: ORIC-114 Dose 3 + amivantamab — ORIC-114 oral daily, amivantamab subcutaneous weekly for 4 weeks followed by every 4 week injection
  Arms: Part 1 Dose Escalation level 3; Part 2 Dose Expansion

SUMMARY:
The purpose of this study is to establish the recommended phase 2 dose (RP2D), safety, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary antitumor activity of ORIC-114 in combination with subcutaneous (SC) amivantamab in patients with advanced or metastatic NSCLC harboring an EGFR exon 20 insertion mutation.

DETAILED DESCRIPTION:
ORIC-114, is a brain penetrant, selective, orally bioavailable, irreversible small molecule inhibitor designed to target EGFR exon 20 insertion mutations, making it a promising therapeutic candidate for development in patients whose tumors harbor these alterations, including those with CNS metastases.

Amivantamab is a bispecific EGFR-directed and MET receptor-directed antibody indicated in combination with carboplatin and pemetrexed for the first line treatment of patients with locally advanced or metastatic NSCLC with EGFR exon 20 insertion mutations and also as a single agent in patients with locally advanced or metastatic NSCLC with EGFR exon 20 insertion mutations whose disease has progressed on or after platinum-based chemotherapy.

This is an open-label, single arm, multicenter, dose escalation followed by dose expansion study to assess the safety and preliminary antitumor activity of ORIC-114 in combination with SC amivantamab, in patients with locally advanced or metastatic NSCLC harboring an EGFR exon 20 insertion mutations.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic NSCLC with a documented EGFR exon 20 insertion mutation as determined locally by any nucleic acid-based diagnostic testing method; all tests should be performed in a CLIA certified or equivalently accredited laboratory
* Prior Therapies:

  1. Dose Escalation: Patients may have previously received and progressed on or after platinum-based chemotherapy or may be treatment naïve
  2. Dose Expansion: Patients must not have received any prior therapy; at time of enrollment, patients must decline, or be ineligible for all available standard of care therapies with proven benefit
* Agreement and ability to undergo a pretreatment biopsy, provided the procedure is clinically feasible and not deemed unsafe by the investigator
* Measurable disease according to RECIST 1.1
* Patients with asymptomatic CNS metastases are eligible
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate organ function

Exclusion Criteria:

* Known small cell lung cancer transformation
* Leptomeningeal disease
* Spinal cord compression not definitively treated with surgery or radiation
* Prior immunotherapy
* Past medical history of interstitial lung disease (ILD), drug induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD
* Active gastrointestinal disease (eg, Crohn's disease, ulcerative colitis, or short gut syndrome) or other malabsorption syndromes that would reasonably impact absorption of ORIC-114

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) | 12 months
  RP2D of ORIC-114 in combination with amivantamab by interval 3+3 dose escalation design
Objective response rate (ORR) | 12 months
  Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Duration of response (DOR) | 12 months
  Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Progression-free survival (PFS) | 12 months
  Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

SECONDARY OUTCOMES:
Plasma PK parameters | 28 Days
  Peak Plasma Concentration (Cmax)
Plasma PK parameters | 28 Days
  Time of maximal plasma concentration (Tmax)
Plasma PK parameters | 28 Days
  Area under the plasma concentration vs time curve (AUC)
Plasma PK parameters | 28 Days
  Apparent plasma terminal elimination half-life (t1/2)
BICR-Objective response rate (ORR) | 12 months
  Blinded independent central review (BICR) according to RECIST 1.1 and RANO-BM
BICR-Duration of response (DOR) | 12 months
  Blinded independent central review (BICR) according to RECIST 1.1 and RANO-BM
BICR-Progression-free survival (PFS) | 12 months
  Blinded independent central review (BICR) according to RECIST 1.1 and RANO-BM
Intracranial Objective response rate (ORR) | 12 months
  Blinded independent central review (BICR) according to RECIST 1.1 and RANO-BM
Intracranial Progression-free survival (PFS) | 12 months
  Blinded independent central review (BICR) according to RECIST 1.1 and RANO-BM

CONTACTS AND LOCATIONS:
Overall Officials: Pratik S. Multani, MD, MS, Study Director — ORIC Pharmaceuticals
Locations (4):
- United States (2):
  - NYU Langone Health, New York, New York
  - Virginia Cancer Specialists, Fairfax, Virginia
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia
- The Princess Margaret Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No